CLINICAL TRIAL: NCT02133755
Title: Effect of Bromocriptine on Insulin Resistance in Polycystic Ovarian Syndrome - A Pilot Study
Acronym: PCOS-Pilot
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Cora fanning, Research Coordinator, IWK Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PCOS-Pilot
Record Dates: First submitted 2014-05-05; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: PCOS; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bromocriptine mesylate (Cycloset) (Other): Cycloset 1.6 to 3.2 mg daily for 3 months
  Interventions: Drug: Bromocriptine

INTERVENTIONS:
Drug: Bromocriptine — Three month administration of bromocriptine. Baseline ultrasound and laboratory parameters measured. Repeat measures at discontinuation of drug at 3 months.
  Other Names: Cycloset

SUMMARY:
The primary aim of this study is to determine the effect of dopamine agonist therapy on insulin resistance in lean vs. obese women with polycystic ovary syndrome. Polycystic ovary syndrome (PCOS) is a common metabolic abnormality in women. The diagnosis of PCOS relies on a constellation of symptoms and signs (problems with ovulation, clinical and/or biochemical signs of hyperandrogenism and cystic ovaries). Though not a diagnostic feature, insulin resistance (IR) is a hallmark of PCOS and up to 80% women with PCOS have IR. Although IR is more significant in obese women with PCOS, even lean women can be insulin resistant. No current therapy addresses the problem of insulin resistance in PCOS. Studies have suggested a dopamine deficiency in patients with PCOS, which may underlie the insulin resistance and may have a pathogenetic role in the development of PCOS. No study to date has assessed the impact of dopamine agonist therapy on IR in patients with PCOS.

DETAILED DESCRIPTION:
Does bromocriptine improve measures of insulin resistance in females with polycystic ovarian syndrome and is there a differential benefit based on Body Mass Index (BMI, kg/m2).

This study will use a single subject design where patients with PCOS will have regular clinical laboratory tests before and after treatment with bromocriptine. It is a pilot study comprised of 20 women with normal BMI (<25) and 40 women with BMI ≥27.

Study data will be collected from participants during regularly scheduled clinic visits (enrolment) and 3 months later (follow-up). Standard care examinations, blood work and pelvic ultrasound will be performed and included as the study data.

The main outcome of interest will be to evaluate the change in HOMA-IR (Homeostatic Model Assessment - Insulin Resistance) from baseline. It is calculated using a fasting glucose and insulin level. Additionally, to determine the magnitude of effect on HOMA-IR as a measure of insulin sensitivity in lean compared to obese women and the effect on insulin sensitivity in those with and without insulin resistance.

Other measure of interest will be a change in glycated hemoglobin (A1C), serum androgens and pituitary hormone levels. No additional tests will be obtained above what is done in the course of usual assessment of patients with PCOS

Change in HOMA-IR values will be calculated for each individual patient and tested using a paired t-test to determine if therapy had a significant impact on HOMA-IR values. A multivariate linear regression will then be applied to determine if this change in HOMA-IR values was influenced by either BMI or baseline HOMA-IR value along with any other potentially confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* women age 18 to 45 years with PCOS willing to maintain consistent weight for 3 month study period

Exclusion Criteria:

* diabetes other conditions associated with insulin resistance previous intolerance to dopamine agonist therapy concomitant medication that would interfere with dopamine agonist therapy insulin resistance syndrome type A or Type B

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Insulin Resistance (IR) | 3 months
  Will bromocriptine improve measures of IR in females with PCOS? IR is a reduced glucose response for given concentration of insulin. IR can be estimated from fasting glucose and insulin levels using the Homeostatic Model Assessment-Insulin Resistance (HOMA-IR) equation: HOMA-IR = fasting plasma glucose (mmol/L) x fasting serum insulin (μU/mL) / 22.5. HOMA-IR correlates well with estimates using the euglycemic clamp method (r = 0.88). A recent study of healthy, young, insulin sensitive, Canadian subjects found that HOMA IR values were 0.78 for Caucasians, 0.82 for East Asians and 1.08 for South Asians. While this demonstrates some ethnic variability, the values for insulin sensitive individuals are lower than traditional cut-off values. With this in mind, and an understanding of the inherent limitations of HOMA-IR, we have chosen a cut-off value of 2, above which we will define insulin resistance and below which, patients will be considered to be insulin sensitive.

SECONDARY OUTCOMES:
IR based on BMI | 3 months
  Is there a differential benefit in insulin resistance reduction based on Body Mass Index (BMI, kg/m2)?

CONTACTS AND LOCATIONS:
Overall Officials: Ali Imran, MD, FRCPC, Principal Investigator — QE II Health Science Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada